CLINICAL TRIAL: NCT03744169
Title: Use of Point-of-care Lung Ultrasound to Diagnose the Etiology of Acute Respiratory Failure in a Pediatric Intensive Care Unit.
Brief Title: Use of Lung Ultrasound to Diagnose the Etiology of Respiratory Failure in a PICU.
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0711; A534285 (Other: UW Madison); SMPH/MEDICINE/PULMON MED (Other: UW Madison); Protocol Version 4/7/2020 (Other: UW Madison)
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Pediatric Respiratory Diseases; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with acute respiratory failure: Point-of-care lung ultrasound on admission to the PICU to determine the cause of respiratory failure.
  Interventions: Diagnostic Test: Lung ultrasound; Diagnostic Test: Clinical exam; Diagnostic Test: Chest x-ray

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — A point-of-care lung ultrasound exam will be performed on admission (no later than 14 hours following admission, allowing for participant stabilization and care) to the PICU and within 6 hours of any escalation in mechanical ventilatory support without interrupting clinical care, by study investigators blinded to participant history, physical examination, and diagnostic testing/imaging and who are not involved in the clinical management of the participant. Investigators will use a six-zone standardized scanning protocol with pattern analysis to form a diagnosis for the cause of the participant's respiratory failure. Images will be acquired by pediatric critical care trainees and saved online; accuracy of diagnoses based on the ultrasound exam will be evaluated by a expert sonographer offline.
Diagnostic Test: Clinical exam — Following morning ICU rounds, the PICU fellow or attending physician caring for the participant will be asked for his/her interpretation of the most recent chest radiograph and his/her diagnosis concerning the etiology of the participant's acute respiratory failure. This clinical diagnosis will be compared to ultrasound findings.
Diagnostic Test: Chest x-ray — Results of chest x-ray will be collected for comparison with ultrasound findings.

SUMMARY:
The purpose of this study is to determine the utility of point-of-care lung ultrasound (POC-LUS) in identifying the etiology of acute respiratory failure in pediatric patients admitted to the pediatric intensive care unit.

DETAILED DESCRIPTION:
Respiratory failure is one of the most common conditions requiring admission to the pediatric intensive care unit (PICU). As such, chest radiography has emerged as the most commonly utilized tool in the assessment of lung pathology despite evidence that it may not be the most accurate. Since the seminal article by Lichtenstein in 2008, lung ultrasound has emerged as an alternative to chest radiography in the assessment of critically ill adults. Likewise, pediatric lung ultrasound has a growing body of research to support its use in commonly encountered lung pathology including pneumonia, asthma, bronchiolitis, acute chest syndrome, pleural effusions, and pneumothorax. Despite the rapidly growing body evidence, there remains little literature to support its use the diagnosis and management of acute respiratory failure in the PICU.

The proposed study will evaluate whether point-of-care lung ultrasound is accurate in determining the etiology of acute respiratory failure on admission to the PICU.

Specific aims include:

* Aim 1: To determine the sensitivity and specificity of point-of-care lung ultrasound examination in identifying the etiology of acute pediatric respiratory failure on admission to the PICU.
* Aim 2: To determine the inter-observer reliability of point-of-care lung ultrasound examination findings in acute pediatric respiratory failure among trainee and expert sonographers.
* Aim 3: Compare point-of-care lung ultrasound with chest radiography in the rate of detection of consolidation, interstitial edema, pneumothorax, and pleural effusion.
* Aim 4: Describe the POC-LUS findings in patients admitted to the PICU with acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 37 weeks gestational age and less than 18 years
* Admitted to PICU
* Clinical diagnosis of acute respiratory failure
* Requirement of non-invasive or invasive respiratory support (as defined by a clinical need for high flow nasal cannula >1L/kg/min; RAM cannula, nasal or full face mask delivered continuous positive airway pressure ventilation; RAM cannula, nasal or full face mask delivered bi-level positive airway pressure ventilation; or invasive mechanical ventilation); requirement of supplemental oxygen with FiO2 > 0.35 while on high flow nasal cannula <1L/kg/min to maintain saturations > 90%; continuous nebulized therapy; or chronic use of home oxygen or ventilator support AND any increase in home settings

Exclusion Criteria:

* Hemodynamically unstable as defined by the initiation of or the need for increased vasopressor support within the previous 30 minutes
* Known chronic respiratory disease such as primary ciliary dyskinesia, cystic fibrosis, or congenital pulmonary malformations.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients age greater than 37 weeks gestational age and less than 18 years old with a clinical diagnosis of acute respiratory failure and the need for non-invasive (HFNC > 1 L/kg/min, CPAP, or BiPAP) or invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity of point-of-care lung ultrasound examination in identifying the etiology of acute pediatric respiratory failure on admission to the PICU | up to one month
  The sensitivity of the lung ultrasound in identifying the etiology of acute pediatric respiratory failure will be determined by comparison with the final criterion or "gold standard" diagnosis generated by a blinded review of the chart after discharge by a study investigator blinded to the case. The hypothesis is that the lung ultrasound performed on admission to the PICU will have a sensitivity of > 90% in determining the etiology of acute respiratory failure in children (as determined by an independent review of the participant's medical record following hospital discharge).
Specificity of point-of-care lung ultrasound examination in identifying the etiology of acute pediatric respiratory failure on admission to the PICU | up to one month
  The specificity of the lung ultrasound in identifying the etiology of acute pediatric respiratory failure will be determined by comparison with the final criterion or "gold standard" diagnosis generated by a blinded review of the chart after discharge by a study investigator blinded to the case. The hypothesis is that the lung ultrasound performed on admission to the PICU will have a specificity of > 90% in determining the etiology of acute respiratory failure in children (as determined by an independent review of the participant's medical record following hospital discharge).

SECONDARY OUTCOMES:
Inter-observer reliability of point-of-care lung ultrasound examination findings in acute pediatric respiratory failure among trainee and expert sonographers | Following acquisition and interpretation of ultrasound images, an average of less than one week
  Ultrasound images obtained by a critical care trainee will be saved online for review by an expert sonographer. The expert sonographer will overread the images; findings will be compared at all ultrasound points to determine percent agreement in interpreting ultrasound exam findings between the trainee and expert sonographer. Additionally final ultrasonographic diagnosis will be compared between trainee and expert sonographers. Interpretation of exam findings and determination of exam diagnosis will be compared to determine the inter-observer reliability of point-of-care lung ultrasound exams in acute pediatric respiratory failure. The hypothesis is that the inter-observer reliability between trainee and expert sonographers for point-of-care lung ultrasound findings will be >80%.

OTHER OUTCOMES:
Rate of pneumothorax detection between point-of-care lung ultrasound and chest radiography | 6 hours before or after completion of chest x-ray
  Chest x-rays findings (as determine by board certified pediatric radiologists) obtained during the course of routine clinical care will be compared to point-of-care lung ultrasound examinations when completed within 6 hours of each other. The hypothesis is that lung ultrasound will have a higher rate of detection of when compared with a chest radiograph taken less than 6 hours prior to or less than 6 hours after lung ultrasound examination.
Rate of pleural effusion detection between point-of-care lung ultrasound and chest radiography | 6 hours before or after completion of chest x-ray
  Chest x-rays findings (as determine by board certified pediatric radiologists) obtained during the course of routine clinical care will be compared to point-of-care lung ultrasound examinations when completed within 6 hours of each other. The hypothesis is that lung ultrasound will have a higher rate of detection of when compared with a chest radiograph taken less than 6 hours prior to or less than 6 hours after lung ultrasound examination.
Rate of interstitial edema detection between point-of-care lung ultrasound and chest radiography | 6 hours before or after completion of chest x-ray
  Chest x-rays findings (as determine by board certified pediatric radiologists) obtained during the course of routine clinical care will be compared to point-of-care lung ultrasound examinations when completed within 6 hours of each other. The hypothesis is that lung ultrasound will have a higher rate of detection of when compared with a chest radiograph taken less than 6 hours prior to or less than 6 hours after lung ultrasound examination.
Rate of alveolar consolidation detection between point-of-care lung ultrasound and chest radiography | 6 hours before or after completion of chest x-ray
  Chest x-rays findings (as determine by board certified pediatric radiologists) obtained during the course of routine clinical care will be compared to point-of-care lung ultrasound examinations when completed within 6 hours of each other. The hypothesis is that lung ultrasound will have a higher rate of detection of when compared with a chest radiograph taken less than 6 hours prior to or less than 6 hours after lung ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Kory, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, American Family Children's Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Namachivayam P, Shann F, Shekerdemian L, Taylor A, van Sloten I, Delzoppo C, Daffey C, Butt W. Three decades of pediatric intensive care: Who was admitted, what happened in intensive care, and what happened afterward. Pediatr Crit Care Med. 2010 Sep;11(5):549-55. doi: 10.1097/PCC.0b013e3181ce7427. PMID 20124947
- [Background] Krmpotic K, Lobos AT. Clinical profile of children requiring early unplanned admission to the PICU. Hosp Pediatr. 2013 Jul;3(3):212-8. doi: 10.1542/hpeds.2012-0081. PMID 24313089
- [Background] Gurney JW. Why chest radiography became routine. Radiology. 1995 Apr;195(1):245-6. doi: 10.1148/radiology.195.1.7892479. No abstract available.
- [Background] Price MB, Grant MJ, Welkie K. Financial impact of elimination of routine chest radiographs in a pediatric intensive care unit. Crit Care Med. 1999 Aug;27(8):1588-93. doi: 10.1097/00003246-199908000-00033. PMID 10470769
- [Background] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718
- [Background] Self WH, Courtney DM, McNaughton CD, Wunderink RG, Kline JA. High discordance of chest x-ray and computed tomography for detection of pulmonary opacities in ED patients: implications for diagnosing pneumonia. Am J Emerg Med. 2013 Feb;31(2):401-5. doi: 10.1016/j.ajem.2012.08.041. Epub 2012 Oct 18. PMID 23083885
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Peris A, Tutino L, Zagli G, Batacchi S, Cianchi G, Spina R, Bonizzoli M, Migliaccio L, Perretta L, Bartolini M, Ban K, Balik M. The use of point-of-care bedside lung ultrasound significantly reduces the number of radiographs and computed tomography scans in critically ill patients. Anesth Analg. 2010 Sep;111(3):687-92. doi: 10.1213/ANE.0b013e3181e7cc42. PMID 20733164
- [Background] Zieleskiewicz L, Cornesse A, Hammad E, Haddam M, Brun C, Vigne C, Meyssignac B, Remacle A, Chaumoitre K, Antonini F, Martin C, Leone M. Implementation of lung ultrasound in polyvalent intensive care unit: Impact on irradiation and medical cost. Anaesth Crit Care Pain Med. 2015 Feb;34(1):41-4. doi: 10.1016/j.accpm.2015.01.002. Epub 2015 Mar 5. PMID 25829314
- [Background] Oks M, Cleven KL, Cardenas-Garcia J, Schaub JA, Koenig S, Cohen RI, Mayo PH, Narasimhan M. The effect of point-of-care ultrasonography on imaging studies in the medical ICU: a comparative study. Chest. 2014 Dec;146(6):1574-1577. doi: 10.1378/chest.14-0728. PMID 25144593
- [Background] Inglis AJ, Nalos M, Sue KH, Hruby J, Campbell DM, Braham RM, Orde SR. Bedside lung ultrasound, mobile radiography and physical examination: a comparative analysis of diagnostic tools in the critically ill. Crit Care Resusc. 2016 Jun;18(2):124. PMID 27242110
- [Background] Expert Round Table on Ultrasound in ICU. International expert statement on training standards for critical care ultrasonography. Intensive Care Med. 2011 Jul;37(7):1077-83. doi: 10.1007/s00134-011-2246-9. Epub 2011 May 26. PMID 21614639
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Frankel HL, Kirkpatrick AW, Elbarbary M, Blaivas M, Desai H, Evans D, Summerfield DT, Slonim A, Breitkreutz R, Price S, Marik PE, Talmor D, Levitov A. Guidelines for the Appropriate Use of Bedside General and Cardiac Ultrasonography in the Evaluation of Critically Ill Patients-Part I: General Ultrasonography. Crit Care Med. 2015 Nov;43(11):2479-502. doi: 10.1097/CCM.0000000000001216. PMID 26468699
- [Background] Levitov A, Frankel HL, Blaivas M, Kirkpatrick AW, Su E, Evans D, Summerfield DT, Slonim A, Breitkreutz R, Price S, McLaughlin M, Marik PE, Elbarbary M. Guidelines for the Appropriate Use of Bedside General and Cardiac Ultrasonography in the Evaluation of Critically Ill Patients-Part II: Cardiac Ultrasonography. Crit Care Med. 2016 Jun;44(6):1206-27. doi: 10.1097/CCM.0000000000001847. PMID 27182849
- [Background] Neskovic AN, Edvardsen T, Galderisi M, Garbi M, Gullace G, Jurcut R, Dalen H, Hagendorff A, Lancellotti P; European Association of Cardiovascular Imaging Document Reviewers:; Popescu BA, Sicari R, Stefanidis A. Focus cardiac ultrasound: the European Association of Cardiovascular Imaging viewpoint. Eur Heart J Cardiovasc Imaging. 2014 Sep;15(9):956-60. doi: 10.1093/ehjci/jeu081. Epub 2014 May 27. PMID 24866902
- [Background] Via G, Hussain A, Wells M, Reardon R, ElBarbary M, Noble VE, Tsung JW, Neskovic AN, Price S, Oren-Grinberg A, Liteplo A, Cordioli R, Naqvi N, Rola P, Poelaert J, Gulic TG, Sloth E, Labovitz A, Kimura B, Breitkreutz R, Masani N, Bowra J, Talmor D, Guarracino F, Goudie A, Xiaoting W, Chawla R, Galderisi M, Blaivas M, Petrovic T, Storti E, Neri L, Melniker L; International Liaison Committee on Focused Cardiac UltraSound (ILC-FoCUS); International Conference on Focused Cardiac UltraSound (IC-FoCUS). International evidence-based recommendations for focused cardiac ultrasound. J Am Soc Echocardiogr. 2014 Jul;27(7):683.e1-683.e33. doi: 10.1016/j.echo.2014.05.001. PMID 24951446
- [Background] Labovitz AJ, Noble VE, Bierig M, Goldstein SA, Jones R, Kort S, Porter TR, Spencer KT, Tayal VS, Wei K. Focused cardiac ultrasound in the emergent setting: a consensus statement of the American Society of Echocardiography and American College of Emergency Physicians. J Am Soc Echocardiogr. 2010 Dec;23(12):1225-30. doi: 10.1016/j.echo.2010.10.005. PMID 21111923
- [Background] Principi N, Esposito A, Giannitto C, Esposito S. Lung ultrasonography to diagnose community-acquired pneumonia in children. BMC Pulm Med. 2017 Dec 19;17(1):212. doi: 10.1186/s12890-017-0561-9. PMID 29258484
- [Background] Xin H, Li J, Hu HY. Is Lung Ultrasound Useful for Diagnosing Pneumonia in Children?: A Meta-Analysis and Systematic Review. Ultrasound Q. 2018 Mar;34(1):3-10. doi: 10.1097/RUQ.0000000000000330. PMID 29112644
- [Background] Stadler JAM, Andronikou S, Zar HJ. Lung ultrasound for the diagnosis of community-acquired pneumonia in children. Pediatr Radiol. 2017 Oct;47(11):1412-1419. doi: 10.1007/s00247-017-3910-1. Epub 2017 Sep 21. PMID 29043420
- [Background] Man SC, Fufezan O, Sas V, Schnell C. Performance of lung ultrasonography for the diagnosis of communityacquired pneumonia in hospitalized children. Med Ultrason. 2017 May 10;19(3):276-281. doi: 10.11152/mu-1027. PMID 28845493
- [Background] Boursiani C, Tsolia M, Koumanidou C, Malagari A, Vakaki M, Karapostolakis G, Mazioti A, Alexopoulou E. Lung Ultrasound as First-Line Examination for the Diagnosis of Community-Acquired Pneumonia in Children. Pediatr Emerg Care. 2017 Jan;33(1):62-66. doi: 10.1097/PEC.0000000000000969. PMID 28045846
- [Background] Chen IC, Lin MY, Liu YC, Cheng HC, Wu JR, Hsu JH, Dai ZK. The role of transthoracic ultrasonography in predicting the outcome of community-acquired pneumonia in hospitalized children. PLoS One. 2017 Mar 16;12(3):e0173343. doi: 10.1371/journal.pone.0173343. eCollection 2017. PMID 28301494
- [Background] Ambroggio L, Sucharew H, Rattan MS, O'Hara SM, Babcock DS, Clohessy C, Steinhoff MC, Macaluso M, Shah SS, Coley BD. Lung Ultrasonography: A Viable Alternative to Chest Radiography in Children with Suspected Pneumonia? J Pediatr. 2016 Sep;176:93-98.e7. doi: 10.1016/j.jpeds.2016.05.033. Epub 2016 Jun 16. PMID 27318374
- [Background] Varshney T, Mok E, Shapiro AJ, Li P, Dubrovsky AS. Point-of-care lung ultrasound in young children with respiratory tract infections and wheeze. Emerg Med J. 2016 Sep;33(9):603-10. doi: 10.1136/emermed-2015-205302. Epub 2016 Apr 22. PMID 27107052
- [Background] Jones BP, Tay ET, Elikashvili I, Sanders JE, Paul AZ, Nelson BP, Spina LA, Tsung JW. Feasibility and Safety of Substituting Lung Ultrasonography for Chest Radiography When Diagnosing Pneumonia in Children: A Randomized Controlled Trial. Chest. 2016 Jul;150(1):131-8. doi: 10.1016/j.chest.2016.02.643. Epub 2016 Feb 26. PMID 26923626
- [Background] Ianniello S, Piccolo CL, Buquicchio GL, Trinci M, Miele V. First-line diagnosis of paediatric pneumonia in emergency: lung ultrasound (LUS) in addition to chest-X-ray (CXR) and its role in follow-up. Br J Radiol. 2016;89(1061):20150998. doi: 10.1259/bjr.20150998. Epub 2016 Jan 22. PMID 26689098
- [Background] Guerra M, Crichiutti G, Pecile P, Romanello C, Busolini E, Valent F, Rosolen A. Ultrasound detection of pneumonia in febrile children with respiratory distress: a prospective study. Eur J Pediatr. 2016 Feb;175(2):163-70. doi: 10.1007/s00431-015-2611-8. Epub 2015 Aug 19. PMID 26283293
- [Background] Urbankowska E, Krenke K, Drobczynski L, Korczynski P, Urbankowski T, Krawiec M, Kraj G, Brzewski M, Kulus M. Lung ultrasound in the diagnosis and monitoring of community acquired pneumonia in children. Respir Med. 2015 Sep;109(9):1207-12. doi: 10.1016/j.rmed.2015.06.011. Epub 2015 Jun 23. PMID 26138897
- [Background] Ho MC, Ker CR, Hsu JH, Wu JR, Dai ZK, Chen IC. Usefulness of lung ultrasound in the diagnosis of community-acquired pneumonia in children. Pediatr Neonatol. 2015 Feb;56(1):40-5. doi: 10.1016/j.pedneo.2014.03.007. Epub 2014 Jul 15. PMID 25034957
- [Background] Pereda MA, Chavez MA, Hooper-Miele CC, Gilman RH, Steinhoff MC, Ellington LE, Gross M, Price C, Tielsch JM, Checkley W. Lung ultrasound for the diagnosis of pneumonia in children: a meta-analysis. Pediatrics. 2015 Apr;135(4):714-22. doi: 10.1542/peds.2014-2833. Epub 2015 Mar 16. PMID 25780071
- [Background] Don M, Barillari A, Cattarossi L, Copetti R; "Italian-Slovenian Group on Lung Ultrasound for Pediatric Pneumonia". Lung ultrasound for paediatric pneumonia diagnosis: internationally officialized in a near future? Acta Paediatr. 2013 Jan;102(1):6-7. doi: 10.1111/apa.12002. Epub 2012 Sep 13. No abstract available. PMID 22924774
- [Background] Shah VP, Tunik MG, Tsung JW. Prospective evaluation of point-of-care ultrasonography for the diagnosis of pneumonia in children and young adults. JAMA Pediatr. 2013 Feb;167(2):119-25. doi: 10.1001/2013.jamapediatrics.107. PMID 23229753
- [Background] Caiulo VA, Gargani L, Caiulo S, Fisicaro A, Moramarco F, Latini G, Picano E, Mele G. Lung ultrasound characteristics of community-acquired pneumonia in hospitalized children. Pediatr Pulmonol. 2013 Mar;48(3):280-7. doi: 10.1002/ppul.22585. Epub 2012 May 2. PMID 22553150
- [Background] Milliner BHA, Tsung JW. Lung Consolidation Locations for Optimal Lung Ultrasound Scanning in Diagnosing Pediatric Pneumonia. J Ultrasound Med. 2017 Nov;36(11):2325-2328. doi: 10.1002/jum.14272. Epub 2017 Jun 6. PMID 28586113
- [Background] Claes AS, Clapuyt P, Menten R, Michoux N, Dumitriu D. Performance of chest ultrasound in pediatric pneumonia. Eur J Radiol. 2017 Mar;88:82-87. doi: 10.1016/j.ejrad.2016.12.032. Epub 2016 Dec 29. PMID 28189214
- [Background] Reali F, Sferrazza Papa GF, Carlucci P, Fracasso P, Di Marco F, Mandelli M, Soldi S, Riva E, Centanni S. Can lung ultrasound replace chest radiography for the diagnosis of pneumonia in hospitalized children? Respiration. 2014;88(2):112-5. doi: 10.1159/000362692. Epub 2014 Jul 2. PMID 24992951
- [Background] Yilmaz HL, Ozkaya AK, Sari Gokay S, Tolu Kendir O, Senol H. Point-of-care lung ultrasound in children with community acquired pneumonia. Am J Emerg Med. 2017 Jul;35(7):964-969. doi: 10.1016/j.ajem.2017.01.065. Epub 2017 Feb 1. PMID 28202294
- [Background] Dankoff S, Li P, Shapiro AJ, Varshney T, Dubrovsky AS. Point of care lung ultrasound of children with acute asthma exacerbations in the pediatric ED. Am J Emerg Med. 2017 Apr;35(4):615-622. doi: 10.1016/j.ajem.2016.12.057. Epub 2016 Dec 26. PMID 28063721
- [Background] Caiulo VA, Gargani L, Caiulo S, Fisicaro A, Moramarco F, Latini G, Picano E. Lung ultrasound in bronchiolitis: comparison with chest X-ray. Eur J Pediatr. 2011 Nov;170(11):1427-33. doi: 10.1007/s00431-011-1461-2. Epub 2011 Apr 6. PMID 21468639
- [Background] Basile V, Di Mauro A, Scalini E, Comes P, Lofu I, Mostert M, Tafuri S, Manzionna MM. Lung ultrasound: a useful tool in diagnosis and management of bronchiolitis. BMC Pediatr. 2015 May 21;15:63. doi: 10.1186/s12887-015-0380-1. PMID 25993984
- [Background] Kader, M., et al., The utility of lung ultrasound in evaluation ofinfants with suspected bronchiolitis.Egypt J of Rad and Nuc Med, 2016. 47(3): p. 1057.
- [Background] Taveira M, Yousef N, Miatello J, Roy C, Claude C, Boutillier B, Dubois C, Pierre AF, Tissieres P, Durand P. [Can a simple lung ultrasound score predict length of ventilation for infants with severe acute viral bronchiolitis?]. Arch Pediatr. 2018 Feb;25(2):112-117. doi: 10.1016/j.arcped.2017.11.005. Epub 2017 Dec 13. French. PMID 29248322
- [Background] Daswani DD, Shah VP, Avner JR, Manwani DG, Kurian J, Rabiner JE. Accuracy of Point-of-care Lung Ultrasonography for Diagnosis of Acute Chest Syndrome in Pediatric Patients with Sickle Cell Disease and Fever. Acad Emerg Med. 2016 Aug;23(8):932-40. doi: 10.1111/acem.13002. Epub 2016 Aug 1. PMID 27155438
- [Background] Raimondi F, Rodriguez Fanjul J, Aversa S, Chirico G, Yousef N, De Luca D, Corsini I, Dani C, Grappone L, Orfeo L, Migliaro F, Vallone G, Capasso L; Lung Ultrasound in the Crashing Infant (LUCI) Protocol Study Group. Lung Ultrasound for Diagnosing Pneumothorax in the Critically Ill Neonate. J Pediatr. 2016 Aug;175:74-78.e1. doi: 10.1016/j.jpeds.2016.04.018. Epub 2016 May 14. PMID 27189678
- [Background] Cattarossi L, Copetti R, Brusa G, Pintaldi S. Lung Ultrasound Diagnostic Accuracy in Neonatal Pneumothorax. Can Respir J. 2016;2016:6515069. doi: 10.1155/2016/6515069. Epub 2016 May 3. PMID 27445558
- [Background] Ng C, Tsung JW. Point-of-care ultrasound for assisting in needle aspiration of spontaneous pneumothorax in the pediatric ED: a case series. Am J Emerg Med. 2014 May;32(5):488.e3-8. doi: 10.1016/j.ajem.2013.11.011. Epub 2013 Nov 13. PMID 24360316
- [Background] Srinivasan S, Cornell TT. Bedside ultrasound in pediatric critical care: a review. Pediatr Crit Care Med. 2011 Nov;12(6):667-74. doi: 10.1097/PCC.0b013e318223147e. PMID 21666528
- [Background] Nguyen J, Amirnovin R, Ramanathan R, Noori S. The state of point-of-care ultrasonography use and training in neonatal-perinatal medicine and pediatric critical care medicine fellowship programs. J Perinatol. 2016 Nov;36(11):972-976. doi: 10.1038/jp.2016.126. Epub 2016 Aug 11. PMID 27513327
- [Background] Su E, Pustavoitau A. Pediatric critical care ultrasound education: the importance of a common denominator. Pediatr Crit Care Med. 2015 Mar;16(3):292-4. doi: 10.1097/PCC.0000000000000342. No abstract available. PMID 25738928
- [Background] Kornblith AE, van Schaik S, Reynolds T. Useful but not used: pediatric critical care physician views on bedside ultrasound. Pediatr Emerg Care. 2015 Mar;31(3):186-9. doi: 10.1097/PEC.0000000000000376. PMID 25706921
- [Background] Lambert RL, Boker JR, Maffei FA. National survey of bedside ultrasound use in pediatric critical care. Pediatr Crit Care Med. 2011 Nov;12(6):655-9. doi: 10.1097/PCC.0b013e3182266a51. PMID 21725274
- [Background] Conlon TW, Himebauch AS, Fitzgerald JC, Chen AE, Dean AJ, Panebianco N, Darge K, Cohen MS, Greeley WJ, Berg RA, Nishisaki A. Implementation of a pediatric critical care focused bedside ultrasound training program in a large academic PICU. Pediatr Crit Care Med. 2015 Mar;16(3):219-26. doi: 10.1097/PCC.0000000000000340. PMID 25607741
- [Background] Conlon TW, Kantor DB, Su ER, Basu S, Boyer DL, Haileselassie B, Petersen TL, Su F, Nishisaki A. Diagnostic Bedside Ultrasound Program Development in Pediatric Critical Care Medicine: Results of a National Survey. Pediatr Crit Care Med. 2018 Nov;19(11):e561-e568. doi: 10.1097/PCC.0000000000001692. PMID 30113518
- [Background] Su E, Pustavoitau A, Hirshberg EL, Nishisaki A, Conlon T, Kantor DB, Weber MD, Godshall AJ, Burzynski JH, Thompson AE. Establishing intensivist-driven ultrasound at the PICU bedside--it's about time*. Pediatr Crit Care Med. 2014 Sep;15(7):649-52. doi: 10.1097/PCC.0000000000000168. PMID 24977438
- [Background] Brogi E, Bignami E, Sidoti A, Shawar M, Gargani L, Vetrugno L, Volpicelli G, Forfori F. Could the use of bedside lung ultrasound reduce the number of chest x-rays in the intensive care unit? Cardiovasc Ultrasound. 2017 Sep 13;15(1):23. doi: 10.1186/s12947-017-0113-8. PMID 28903756
- [Background] Alpert EA, Amit U, Guranda L, Mahagna R, Grossman SA, Bentancur A. Emergency department point-of-care ultrasonography improves time to pericardiocentesis for clinically significant effusions. Clin Exp Emerg Med. 2017 Sep 30;4(3):128-132. doi: 10.15441/ceem.16.169. eCollection 2017 Sep. PMID 29026885
- [Background] Raman D, Sharma M, Moghekar A, Wang X, Hatipoglu U. Utilization of Thoracic Ultrasound for Confirmation of Central Venous Catheter Placement and Exclusion of Pneumothorax: A Novel Technique in Real-Time Application. J Intensive Care Med. 2019 Jul;34(7):594-598. doi: 10.1177/0885066617705839. Epub 2017 Apr 26. PMID 28443388
- [Background] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127
- [Background] Lichtenstein, D.A. and G.A. Meziere, The BLUE-points: threestandardized points used in the BLUE-protocol for ultrasound assessment of thelung in acute respiratory failure.Critical Ultrasound Journal, 2011. 3(2): p. 109-110.
- [Derived] DeSanti RL, Al-Subu AM, Cowan EA, Kamps NN, Lasarev MR, Schmidt J, Kory PD. Point-of-Care Lung Ultrasound to Diagnose the Etiology of Acute Respiratory Failure at Admission to the PICU. Pediatr Crit Care Med. 2021 Aug 1;22(8):722-732. doi: 10.1097/PCC.0000000000002716. PMID 33739956